CLINICAL TRIAL: NCT05491057
Title: A Multicenter, Open-label, Single-arm, Non-interventional Study to Investigate the Treatment Patterns of Nerlynx® (Neratinib) in HER2-positive Early-stage Breast Cancer in China
Brief Title: Treatment Patterns of Neratinib in HER2+ EBC in China
Status: Not yet recruiting | Type: Observational
Sponsor: Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Other Study IDs: PF008
Record Dates: First submitted 2022-07-27; First posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — neratinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Neratinib extended ajuvant treatmeng for 1 year
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — Neratinib standard dose 240 mg once daily for 1 year

SUMMARY:
This is a multicenter, open-label, single-arm, non-interventional study to investigate the treatment patterns of Neratinib in HER2-positive early-stage breast cancer in China

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent approved by the reviewing Ethics Committee (EC).
* Adult patients (≥18 years of age, no upper limit).
* Eligible to receive neratinib for extended adjuvant treatment as per prescribing information in China, diagnosed with HER2 overexpressing/amplified early-stage breast cancer regardless of hormone receptor (HR) status and clinical/radiological assessed to be negative for recurrences or metastatic disease.

Exclusion Criteria:

* Presence of any contraindication with regard to the neratinib treatment.
* Current or upcoming participation in an interventional clinical trial. (Investigational treatment within four weeks of enrolment).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients assigned extended adjuvant treatment with neratinib for 12 months for their HER2-positive, early-stage breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Duration of Treatment | 12 months of treatment
  Median duration of extended adjuvant treatment with neratinib
Treatment holds and permanent discontinuations time | 12 months of treatment
  Median treatment holds and permanent discontinuations time

SECONDARY OUTCOMES:
Patient demographics | Baseline
  % of patients with different demographic characteristics
Patient characteristics | Baseline
  % of patients with different disease characteristics
Time to treatment | Baseline
  Median time to treatment since completion of adjuvant regimen
Prior adjuvant treatments | Baseline
  % of patients with different prior adjuvant treatments
Dose adjustments | 12 months of treatment
  % of patients with dose adjustments
Dose intensity | 12 months of treatment
  Absolute and relative dose intensity
Concomitant medication | 12 months of treatment
  % of patients with different concomitant medications
Incidence of AESI | 12 months of treatment
  Incidence of all grades of adverse events of special interest (AESI)
Type of AESI | 12 months of treatment
  % of different type of all grades of adverse events of special interest (AESI)
Severity of AESI | 12 months of treatment
  % of patients with adverse events by severity
action taken for AESI | 12 months of treatment
  % of patients with action taken against adverse events

OTHER OUTCOMES:
Time of recurrence | 12 months of treatment； 12 months of follow-up
  Time from end of neratinib treatment to first invasive recurrence
Recurrent site | 12 months of treatment； 12 months of follow-up
  % of different site of invasive tumor recurrence
Recurrent size | 12 months of treatment； 12 months of follow-up
  % of different size of invasive tumor recurrence
QoL - EQ-5D-5L | 12 months of treatment
  Median score of the EQ-5D-5L during neratinib treatment. EQ-5D-5L scale as self-reported health-related quality of life.
QoL - FACIT D | 12 months of treatment
  Median score of the FACIT D during neratinib treatment. FACIT D scale as self-reported health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Affair, Shanghai, China

IPD SHARING:
Plan to Share IPD: No